CLINICAL TRIAL: NCT05351944
Title: Dialectical Behavioral Therapy Skills for Impulsive Aggression in Children Diagnosed with Attention Deficit Hyperactivity Disorder At Alexandria University Hospitals
Brief Title: Dialectical Behavioral Therapy Skills for Impulsive Aggression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Aya Maged, Doctor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 850486055
Record Dates: First submitted 2022-04-19; First posted 2022-04-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Impulsive Aggression; ADHD; Executive Dysfunction
Keywords: DBT; aggression; ADHD; biomarkers; executive functions
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Aggression | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Randomized control clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The intervention group (group A) DBT skills (Experimental): Will attend Dialectical Behavioral Therapy skills group for both the children and their parents, DBT is an evidence based comprehensive cognitive behavioral treatment for complex mental disorders and have been adapted for intractable behavioral disorders involving emotion dysregulation, skills will be provided in group therapy as fixed weekly sessions over 9-month duration for all the children and the parents in group A including:
  1. Emotion regulation skills module over 8 weeks.
  2. Mindfulness skills module over 3 weeks
  3. Interpersonal effectiveness skills module over 7 weeks.
  4. Distress tolerance skills module over 8 weeks.
  5. Walking the middle path skills module over 3 weeks.
  Interventions: Behavioral: Dialectical behavioral therapy skills for the intervention experimental group A
- the control group (group B) (Active Comparator): Will receive psychoeducation and medications targeting ADHD symptoms (stimulants or atomoxetine according to FDA approved dose per age and weight) according to the international guidelines for management of ADHD according to symptom severity, given that assessment before and after intervention will be done by different medical personnel than those providing the intervention for the two groups.
  Interventions: Drug: psychoeducation or Atomoxetine or stimulants according to ADHD severity

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy skills for the intervention experimental group A — Our hypothesis is that impulsive aggression as evidenced by inflammatory biomarkers might improve by targeting executive dysfunctions with Dialectical Behavioural Therapy skills modules directed to the children and their parents in the form of response inhibition dysfunctions with Dialectical Behavioural Therapy mindfulness and distress tolerance skills modules, emotion regulation executive dysfunctions with Dialectical Behavioural Therapy emotion regulation skills module and socioenvironmental factors with interpersonal effectiveness and walking the middle path Dialectical behavioural therapy skills modules.
  Arms: The intervention group (group A) DBT skills
Drug: psychoeducation or Atomoxetine or stimulants according to ADHD severity — the control group (group B) will receive psychoeducation and medications targeting ADHD symptoms (Atomoxetine or stimulants according to FDA approved dose according to age and weight ) according to the international guidelines for management of ADHD according to symptom severity
  Arms: the control group (group B)

SUMMARY:
This trial aims to Study the efficacy of DBT skills for impulsive aggression and executive dysfunctions in drug naïve children who are presented with impulsive aggression and ADHD and attending Child and adolescent clinic at Alexandria university hospitals using weekly group therapy for 8 month and testing pre and posttreatment biomarkers of aggression.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 6 to 13-year-old.
* Patients diagnosed with ADHD and presented with impulsive aggression.
* Commitment to therapy from the child and the parent.
* Written consent of all the children parents.
* Male gender.
* Drug naïve or stopped medications for at least one month.

Exclusion Criteria:

* Patients younger than 6 years of age as it's the starting age for DBT-C.
* Patients who dropped from DBT skills group (missing more than 3 consecutive sessions) whether the child or his parent.
* Patients diagnosed with drug abuse.
* Patients with severe sensory impairment or intellectual disability.
* Drug induced aggression as levetiracetam, topiramate and benzodiazepines.
* Patients diagnosed with Autism spectrum disorder or psychotic disorders.

Ages: 6 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-05-07 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Impulsive aggression severity | Change from Baseline at 12 month
  Using Modified overt aggression scale ,This scale rates the patient's aggressive behavior regarding four types of aggression (verbal, against objects, against self, against others) to give a total MOAS score about the patient's aggressive behavior. Each type of aggression had a rating of 0 when aggression was absent and four levels of severity. Weighted scores are then added together to yield the total score.
Biomarkers of aggression 1 | Change from Baseline 12 month
  quantitative CRP
Biomarkers of aggression 2 | Change from Baseline 12 month
  interleukin 6
Biomarkers of aggression 3 | Change from Baseline 12 month
  Serum cortisol level (at 9 am and 9 pm) using The enzyme-linked immunosorbent assay (ELISA) technique

SECONDARY OUTCOMES:
Executive dysfunctions severity | Change from Baseline 12 month
  using Barkley Deficits In Executive Functioning Scale - Children and Adolescents ,The manuals indicate that results from the scale can be interpreted using normative comparisons (percentile scores based on sex and age group
ADHD symptom severity | Change from Baseline 12 month
  using Conner's parent rating scale for ADHD pre and post treatment to assess change in severity

CONTACTS AND LOCATIONS:
Overall Officials: aya maged, master, Principal Investigator — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No